CLINICAL TRIAL: NCT01539954
Title: Computerized Alcohol Screening for Children and Adolescents (cASCA) in Primary Care
Brief Title: Computerized Alcohol Screening for Children and Adolescents
Acronym: cASCA
Status: Withdrawn | Type: Observational
Why Stopped: The project was not funded.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Other Study IDs: JK_NIAAA_02-12
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Related Disorders
Keywords: Alcohol related disorders
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Youth 9-18 years of age

SUMMARY:
The goal of this project is to develop a computerized screening program for primary care offices that is based on the NIAAA's Alcohol Screening Guide for Children and Adolescents and assess its psychometric properties among nine- to 18-yr-old primary care patients. There have been few studies of alcohol screening and brief intervention conducted among adolescents receiving primary medical care. This project will develop and validate a new computerized Alcohol Screening for Children and Adolescents (cASCA) system based on the two age-specific screening questions of the NIAAA Guide and includes the CRAFFT and AUDIT as secondary risk and problem assessments. The system will yield a provider report with the screening results, level of risk, and recommended brief advice, counseling, or referral strategies. The Specific Aims of this project are to: 1)Assess the sensitivity, specificity, positive and negative predictive values of the 'any drinking/number of drinking days' and 'friends' questions of the cASCA in identifying past-year use as determined by the Timeline Follow-Back Calendar (TLFB), and for identifying any problem use, abuse or dependence as determined by the AUDIT, CRAFFT and a structured psychiatric diagnostic interview (computerized DISC-IV, Youth Version) at baseline (criterion validity); 2)Assess the test-retest reliability of the cASCA in measuring drinking frequency categories and in classifying patients into Low, Medium and High risk categories; 3)Assess the predictive validity of the 'any drinking/number of drinking days' and 'friends' questions in predicting drinking, "binge" drinking, and any problem use, abuse or dependence at 12-mos follow-up; 4)Assess the degree to which the 'any drinking/number of drinking days' item of the cASCA predicts drug use risk as measured by the TLFB (any use and frequency), tobacco use as measured by the Hooked on Nicotine Checklist (screen for potential nicotine dependence), drug use disorders as measured by the Drug Abuse Screening Test for Adolescents, and the degree to which it predicts other mental health problems as measured by the Youth DISC Predictive Scales at baseline and 12-month follow-up; 5)Compare the psychometric properties of the cASCA across subgroups, including: age, gender, race/ethnicity, practice type, provider type, and patient risks (e.g., those with/without friends who drink); and explore the possible effects of the cASCA system on drinking at 3-, 6-, 9-, and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* nine- to 18-years old
* arriving for non-emergent care
* have an email address and internet access
* provide informed assent/consent.

Exclusion Criteria:

* unable to read or understand English
* living away at college at the time of the recruitment visit
* not available for computer/telephone follow-ups
* judged by the provider to be medically or emotionally unstable at time of visit.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth 9-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensitivity of cASCA | Baseline
  We will examine validity of the lifetime "any drinking" item by comparing participant responses on the c-ASCA to responses on the Brief Substance Use History (BSUH) questionnaire (lifetime use and age of initiation of use, if any).

SECONDARY OUTCOMES:
Test-retest reliability of cASCA | baseline
  We will calculate Cohen's kappas to evaluate 1-2 week test-retest agreement on c-ASCA responses
Validity of "number of drinking days" item in c-ASCA | Baseline
  For middle and high school-aged youth (12-18 yrs), we will examine validity of the c-ASCA past-year "number of drinking days" by computing the intra-class correlation coefficients (ICC) assessing agreement between the two continuous variables of total past-year number of days reported on c-ASCA and on the TLFB.

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Adolescent Substance Abuse Research — http://www.ceasar.org